CLINICAL TRIAL: NCT00562757
Title: The Harbinger ICD Patient (HIP) Study
Brief Title: Prospective Study to Identify Patients at Risk of Dangerous Ventricular Arrhythmias
Acronym: HIP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Harbinger Medical, Inc. (Industry)
Other Study IDs: HMI-HIP
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Sudden Cardiac Death
Keywords: Wedensky modulation; Risk stratification; Electrophysiology; Noninvasive; Ischemic heart disease; ICD guidelines; Myocardial infarction
MeSH Terms: conditions — Death, Sudden, Cardiac; Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Post myocardial infarction patients who received an ICD, stratified into low versus high WMI groups

SUMMARY:
The purpose of this study is to determine how well the device predicts susceptability to potentially lethal ventricular arrhythmias.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) accounts for half of all deaths from cardiovascular causes, with an annual incidence of 1 to 2 deaths per 1000 population. In the United States this translates to between 300,000 to more than 400,000 deaths annually. Results from numerous large, well designed clinical trials have demonstrated the efficacy of the implantable cardioverter-defibrillator (ICD) for improving survival in patients with ischemic heart disease. However, measures used to risk stratify patients, such as left ventricular ejection fraction do not adequately identify those patients who can most benefit from ICD therapy. As a result, many patients who currently receive an ICD do not use the device. In addition, many more patients who could benefit from ICD therapy are outside of current guidelines and do not have access to this life-saving therapy.

This prospective study was intended to determine how well the Harbinger Wedensky Modulation Index (WMI) technique risk stratifies patients into two groups: those needing antiarrhythmic therapy and those who do not need antiarrhythmic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Post myocardial infarction patients receiving ICD therapy

Exclusion Criteria:

* Patients unable to give consent
* Pacemaker dependant patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post myocardial infarction patients who received an ICD are included. Enrollment is at eight sites - four in the USA and four in three European countries. The enrollment sites are hospitals and teaching institutions.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2003-09; Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Life Threatening Cardiac Event (death or annotated malignant ventricular arrhythmia detected by ICD and confirmed by cardiologist review) | Up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Harold Hoium, MBA, Study Director — Harbinger Medical, Inc.
Locations (8):
- United States (4):
  - Arizona Arrhythmia Consultants, Phoenix, Arizona
  - Galichia Heart Hospital, Wichita, Kansas
  - Caritas St. Elizabeth's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
- Germany (2):
  - University of Bonn, Bonn
  - University of Mannheim, Mannheim
- Rikshospital, Oslo, Norway
- Kantonsspital Luzern, Lucerne, Switzerland